CLINICAL TRIAL: NCT05208216
Title: Electronic Neuromuscular Stimulation Versus Intermittent pneumAtic Compression Devices for the pRevention of Venous Thromboembolic Disease in Critically Ill Adults: a Randomised Feasibility Study
Brief Title: Neuromuscular Stimulation Versus Intermittent Compression for Venous Thromboembolism Prophylaxis in Critical Care
Acronym: ENSARIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Firstkind Ltd (Industry); Manchester Academic Health Science Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B01316
Record Dates: First submitted 2021-12-13; First posted 2022-01-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; Sepsis; Acute Illness; Venous Thromboembolism
Keywords: venous thromboembolism; Critical illness
MeSH Terms: conditions — Critical Illness; Sepsis; Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Application of the Geko device for mechanical VTE prophylaxis up until day 10 / discharge form critical care (whichever comes sooner).
  Interventions: Device: Geko device
- Usual care arm (Active Comparator): Application of our usual intermittent pneumatic compression devices for mechanical VTE prophylaxis up until day 10 / discharge form critical care (whichever comes sooner).
  Interventions: Device: Flowtron DVT

INTERVENTIONS:
Device: Geko device — A small battery powered device that provides neuromuscular stimulation to the muscles of the lower leg to enhance venous return from the leg and reduce the risk of patient developing VTE.
  Arms: Intervention arm
Device: Flowtron DVT — A pneumatically powered pair of calf boots device that intermittently compress the muscles of the lower leg to enhance venous return from the leg and reduce the risk of patient developing VTE.
  Arms: Usual care arm

SUMMARY:
In this prospective, randomised, open-label, parallel group, feasibility trial; the investigators will objectively assess whether it is feasible to apply the Geko device to critically ill adults for the prevention of venous thromboembolism (VTE) compared to usual care with intermittent pneumatic compression devices (IPCs).

DETAILED DESCRIPTION:
VTE is a common problem amongst patients in critical care. Current measures include intermittent pneumatic compression devices, used to aid the venous return of blood from the lower limbs. These devices are contraindicated and/or poorly tolerated by some patients. Neuromuscular stimulation of the lower leg muscles might offer a better tolerated and more physiological alternative to IPCs.

In this feasibility trial the investigators will randomly allocate 40 patients to receive either the Geko device (n=20) or IPCs (n=20) as principal means of mechanical VTE prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 18 years.
* Intact healthy skin at the proposed site of gekoTM device application.
* Within 24 hours of their admission to critical care
* Expected to remain in critical care until the day after tomorrow

Exclusion Criteria:

* Use of any concurrent neuro-modulation drug or device (e.g. neuromuscular blocking agents).
* Trauma to the lower limbs that would prevent geko™ from stimulating the common peroneal nerve.
* Inability to palpate the fibula head in order to apply geko device effectively
* Inability to obtain valid written consent from the participant or their designated legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Successful application of the intervention | Daily measurements up to day 10 after enrolment
  Objective measures of feasibility will include successful application of the intervention device. Investigators will make a daily assessment of whether the device is successfully applied to a participant or not. Successful application is defined as a device applied and producing a visible muscle twitch in the participant's lower leg. A predefined threshold of 70% or above would indicate feasibility of effective application of the intervention to trial participants.

SECONDARY OUTCOMES:
Venous return in the lower limbs | Baseline & day 3-5.
  Objective measurements of blood velocity in the femoral veins will be made through expert bedside ultrasound scans on participant's lower limbs. Two assessments of this outcome will be made, one at baseline prior to application of any device and another between days 3-5.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester Royal Infirmary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Geko Device Homepage — https://www.gekodevices.com/